CLINICAL TRIAL: NCT06777108
Title: Pharmacokinetics of Berkeley Life Oral Nitrate Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Arthur L Weltman, Professor of Kinesiology, University of Virginia
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HSR230481
Record Dates: First submitted 2025-01-03; First posted 2025-01-15 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-01

CONDITIONS: Hypertension
Keywords: Nitric Oxide; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Participants will take a single-dose (two capsules) of the Berkeley Life Pro supplement. Saliva and blood will be assessed at multiple timepoints: baseline, 2 hours, 4 hours, 8 hours, and 24 hours following supplementation. Participants will then have the option to participate in a second crossover supplementation protocol following at least a one-week washout period where they will take a ½ dose (one capsule) of the Berkeley Life Pro supplement. Saliva and blood will be assessed at multiple timepoints: baseline, 2 hours, 4 hours, 8 hours, and 24 hours following supplementation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single Dose - Two Capsules (Experimental): Participants will take a single-dose (two capsules) of the Berkeley Life Pro supplement. Saliva and blood will be assessed at multiple timepoints: baseline, 2 hours, 4 hours, 8 hours, and 24 hours following supplementation.
  Interventions: Dietary Supplement: Inorganic Nitrate
- 1/2 Dose - Single Capsule (Experimental): Participants will have the option to participate in a second supplementation protocol following at least a one-week washout period where they will take a ½ dose (one capsule) of the Berkeley Life Pro supplement. Saliva and blood will be assessed at multiple timepoints: baseline, 2 hours, 4 hours, 8 hours, and 24 hours following supplementation.
  Interventions: Dietary Supplement: Inorganic Nitrate

INTERVENTIONS:
Dietary Supplement: Inorganic Nitrate — The intervention evaluates the single and 1/2-dose pharmacokinetics of a plant-based bioequivalent inorganic nitrate (NO3-) complex with vitamins, antioxidantsand phytophenol rich food extracts.
  Other Names: Berkeley Life Pro Capsules

SUMMARY:
The purpose of the study is to examine the way that a nitric oxide supplement moves through the body. Specifically, the relationship between saliva and blood concentration of the supplement and the elapsed time since taking the supplement.

Participants will :

* Come to UVA to participate in testing procedures.
* Take a nitric oxide supplement up to twice.
* Complete a pregnancy test if the participant is a pre-menopausal female.
* Produce saliva into a tube to collect a sample.
* Undergo several blood draws (less than 6 tablespoons).
* Wear a 24-hour non-invasive device that monitors the participant's blood pressure.

DETAILED DESCRIPTION:
Nitric oxide (NO) is a gaseous, diatomic free-radical that is essential for a variety of physiological functions, including tissue perfusion, mitochondrial function, and glucose regulation. Patients with cardiovascular disease (CVD) are often marked by decreased NO bioavailability due to disruptions in the endothelium through a variety of CVD risk factors including hypertension, diabetes, and inflammation. Recently, an alternative exogenous route to increase NO bioavailability in patients with CVD has been explored via oral supplementation of inorganic nitrate (NO3-) and the subsequent elevation of plasma nitrite (NO2-). This approach has been applied across a range of human healthy and clinical conditions. Several comprehensive reviews on the role of nitrate in cardiovascular health have been published, and there have been more than 60 randomized controlled trials (RCTs) investigating the effects of dietary nitrate from plant sources on markers of cardiovascular health (blood pressure, endothelial function, arterial stiffness, platelet reactivity and platelet aggregation).

There is a consensus on the principal pathways and primary mechanisms involved in the conversion of oral NO3- to circulating NO2- and NO, however, there remains significant variation in the levels of NO metabolites attained in the plasma that is dependent upon the type of oral inorganic nitrate supplementation. Reduction of inorganic nitrate to bioavailable NO is a two-cycle process:

1. Inorganic nitrate is swallowed and absorbed into the circulation, where a proportion is then sequestered and concentrated in the salivary glands and slowly released into the oral cavity. At this stage commensal bacteria reduce nitrate to nitrite in the oral cavity;
2. Nitrite is swallowed and absorbed into the circulation. This circulating nitrite is readily reduced to nitric oxide by a variety of pathways involving single-electron transfer reactions with protons (H+) and hemeproteins (i.e., hemoglobin, myoglobin) during deoxygenation.

Given the dearth of other ways in human physiology to reduce nitrate to nitrite this process is highly reliant on the bacterial species within the oral microbiome. The investigators of this study (and others) have also shown that disruption of the oral microbiome via commercially available anti-bacterial mouthwash abolished increases in plasma nitrite following oral inorganic nitrate supplementation (in the form of beetroot juice) and blunted reductions in blood pressure, compared to placebo control conditions. Additionally, the investigators of this study have also shown that circulating levels of nitrite in healthy volunteers were higher compared with patients with diabetes and/or peripheral artery disease.

The potential for reduced endogenous NO and associated circulating plasma NO2- in populations at risk for cardiovascular disease (older, hypertensive, obese) make the exogenous pathway of oral supplementation and bacterial reduction of NO3- to NO2- (and subsequently NO), a potentially novel therapeutic approach to increase vascular health.

The purpose of the current proposal is to examine the single dose pharmacokinetics (the relationship between supplement plasma concentration and the time elapsed since the supplement's administration) of "Berkeley Life Pro Capsules" (Chicago, IL). Specifically, plasma and salivary nitrate and nitrite concentrations will be collected and measured at baseline (0) and 2, 4, 8 and 24 hours following two different doses of "Berkeley Life Pro Capsules" 314mg inorganic nitrate (2 capsules) (n=12) and 167mg inorganic nitrate (1 capsule) (n=6).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to communicate meaningfully with the investigator and must be legally competent to provide written informed consent.
* Subjects may be of either sex with age ≥ 18 years
* Blood pressure >120 systolic and >80 diastolic at rest

Exclusion Criteria:

* Significant cardiac or other medical history
* Medication changes within the previous six months
* Oral antibiotic use within previous four weeks
* Oral cancer/severe oral disease
* Using an over-the-counter antibacterial mouthwash or a mouthwash containing chlorhexidine and unwilling to discontinue use
* Use of a prescription chlorhexidine or antibacterial mouthwash.
* Current tobacco users
* Pregnant or lactating females
* Currently taking nitroglycerine (or other inorganic nitrates), PDE-5 inhibitors (ex: Cialis, Viagra), or xanthine oxidase inhibitors (ex: Allopurinol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-04-06 (Actual); Study Completion 2024-04-06 (Actual)

PRIMARY OUTCOMES:
Change in plasma nitrite | 24-hours following supplementation (data collected at baseline (before supplementation), 2 hours, 4 hours, 8 hours, and 24 hours following supplementation.
  Change in plasma nitrite over a 24-hour period. Measured at the following timepoints: baseline (before single-dose supplementation), 2 hours, 4 hours, 8 hours, and 24 hours following single-dose supplementation.

SECONDARY OUTCOMES:
Change in plasma nitrate | 24-hours following supplementation (data collected at baseline (before supplementation), 2 hours, 4 hours, 8 hours, and 24 hours following supplementation.
  Change in plasma nitrate over a 24-hour period. Measured at the following timepoints: baseline (before single-dose supplementation), 2 hours, 4 hours, 8 hours, and 24 hours following single-dose supplementation.

OTHER OUTCOMES:
Change in saliva nitrite | 24-hours following supplementation (data collected at baseline (before supplementation), 2 hours, 4 hours, 8 hours, and 24 hours following supplementation.
  Change in saliva nitrite over a 24-hour period. Measured at the following timepoints: baseline (before supplementation), 2 hours, 4 hours, 8 hours, and 24 hours following supplementation.
Change in saliva nitrate | 24-hours following supplementation (data collected at baseline (before supplementation), 2 hours, 4 hours, 8 hours, and 24 hours following supplementation.
  Change in saliva nitrate over a 24-hour period. Measured at the following timepoints: baseline (before single-dose supplementation), 2 hours, 4 hours, 8 hours, and 24 hours following single-dose supplementation.
Changes in 24-hour blood pressure | 24-hour period following supplementation (data collected every 30 minutes)
  Changes in blood pressure during the 24-hour period following supplementation.
Difference in plasma nitrate changes between single dose and 1/2 dose of supplement | 24-hours following each supplementation type (single dose and 1/2 dose) (data collected at baseline (before supplementation, 2 hours, 4 hours, 8 hours, and 24 hours post-supplementation)
  Differences in plasma nitrate changes at each timepoint between a single capsule and two capsules. Measured at the following timepoints: baseline (before single-dose supplementation and 1/2 dose supplementation), 2 hours, 4 hours, 8 hours, and 24 hours following single-dose supplementation and 1/2 dose supplementation.
Difference in plasma nitrite changes between single dose and 1/2 dose of supplement | 24-hours following each supplementation type (single dose and 1/2 dose) (data collected at baseline (before supplementation, 2 hours, 4 hours, 8 hours, and 24 hours post-supplementation)
  Differences in plasma nitrite changes at each timepoint between a single capsule and two capsules. Measured at the following timepoints: baseline (before single-dose supplementation and 1/2 dose supplementation), 2 hours, 4 hours, 8 hours, and 24 hours following single-dose supplementation and 1/2 dose supplementation.
Difference in saliva nitrate changes between single dose and 1/2 dose of supplement | 24-hours following each supplementation type (single dose and 1/2 dose) (data collected at baseline (before supplementation, 2 hours, 4 hours, 8 hours, and 24 hours post-supplementation)
  Differences in saliva nitrate changes at each timepoint between a single capsule and two capsules. Measured at the following timepoints: baseline (before single-dose supplementation and 1/2 dose supplementation), 2 hours, 4 hours, 8 hours, and 24 hours following single-dose supplementation and 1/2 dose supplementation.
Difference in saliva nitrite changes between single dose and 1/2 dose of supplement | 24-hours following each supplementation type (single dose and 1/2 dose) (data collected at baseline (before supplementation, 2 hours, 4 hours, 8 hours, and 24 hours post-supplementation)
  Differences in saliva nitrite changes at each timepoint between a single capsule and two capsules. Measured at the following timepoints: baseline (before single-dose supplementation and 1/2 dose supplementation), 2 hours, 4 hours, 8 hours, and 24 hours following single-dose supplementation and 1/2 dose supplementation.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia Student Health and Wellness Buidling, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No